CLINICAL TRIAL: NCT04750070
Title: Randomized Controlled Trial of Dopamine, Adrenaline, and Blood Transfusion for Treatment of Fluid Refractory Shock in Children With Severe Acute Malnutrition or Severe Underweight and Cholera or Other Dehydrating Diarrheas
Brief Title: Management of Shock in Children With SAM or Severe Underweight and Diarrhea
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of British Columbia (Other); Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-20021
Record Dates: First submitted 2021-02-01; First posted 2021-02-11 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Shock Hypovolemic; Shock, Septic; Blood Transfusion; Adrenaline; Dopamine
Keywords: Severe acute malnutrition; Children; Shock; Cholera; Dehydrating diarrhea; Severe underweight; Acute malnutrition
MeSH Terms: conditions — Shock; Shock, Septic; Severe Acute Malnutrition; Cholera; Thinness | interventions — Blood Specimen Collection; Dopamine; Epinephrine

STUDY DESIGN:
Intervention Model Description: Systematic evaluation of the effects of blood transfusion and inotrope(s) and vasopressor in children with dehydrating diarrhea (for example, in cholera) and acute malnutrition having fluid refractory shock and unresponsive to WHO standard fluid therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blood Transfusion and Dopamine arm (Active Comparator): Children in this group (Treatment plan A) will receive a transfusion of whole human blood in a dose of 10 mL/kg over 2-3 hours. In addition, they will receive dopamine, 8 microgram/kg/min (increasing the dose after 15 minutes to 12 microgram/kg/min to a maximum of 15 microgram/kg/min)
  Interventions: Drug: Blood and Dopamine
- Blood Transfusion and Adrenaline arm (Experimental): Children in this group (Treatment plan B) will receive a transfusion of whole human blood in a dose of 10 mL/kg over 2-3 hours. In addition, they will receive adrenaline, 0.1 microgram/kg/min (increasing the dose after 15 minutes to 0.2 microgram/kg.min to a maximum of 0.3 microgram/kg.min)
  Interventions: Drug: Blood and adrenaline

INTERVENTIONS:
Drug: Blood and Dopamine — Children in this group will receive a transfusion of whole human blood in a dose of 10 mL/kg over 2-3 hours. They will also receive dopamine, 8 microgram/kg.min (increasing the dose after 15 minutes to 12 microgram/kg/min to a maximum of 15 microgram/kg/min)
  Other Names: Dopamine; Blood
  Arms: Blood Transfusion and Dopamine arm
Drug: Blood and adrenaline — Children in this group will receive a transfusion of whole human blood in a dose of 10 mL/kg over 2-3 hours. They will also receive adrenaline, 0.1 microgram/kg/min (increasing the dose after 15 minutes to 0.2 microgram/kg.min to a maximum of 0.3 microgram/kg.min)
  Other Names: Epinephrine; Blood
  Arms: Blood Transfusion and Adrenaline arm

SUMMARY:
Diarrhea is one of the leading causes of under-five childhood mortality and accounts for 8% of 5.4 million global under-5 deaths. The coexistence of sepsis and hypovolemic shock in children with severe acute malnutrition (SAM) having diarrhea is common. At Dhaka hospital of icddr,b, the death rate is as high as 40% and 69% in children with severe sepsis and septic shock respectively with co-morbidities such as severe malnutrition.

The conventional management of SAM children with features of severe sepsis recommended by WHO includes administration of boluses of isotonic saline followed by blood transfusion in unresponsive cases with septic shock; whereas the Surviving Sepsis Campaign (SSC) guideline recommends vasoactive support. To date, no study has evaluated systematically the effects of inotrope(s) and vasopressor or blood transfusion in children with dehydrating diarrhea (for example, in cholera) and SAM having shock and unresponsive to WHO standard fluid therapy.

This randomized trial will generate evidence whether inotrope and vasopressor or blood transfusion should be selected for severely malnourished children having hypotensive shock and who failed to respond to WHO standard fluid bolus.

DETAILED DESCRIPTION:
Background:

1. Burden: Burden: Diarrhea is one of the leading causes of under-five childhood mortality and accounts for 8% of 5.4 million global under-5 deaths. Co-morbidity of severe acute malnutrition (SAM) and shock in children with diarrhea is associated with increased mortality. Nearly half of the patients admitted to the Intensive Care Unit (ICU) of Dhaka Hospital of icddr,b present with sepsis. Data demonstrates that about 43% of children progressed from severe sepsis to septic shock despite receiving recommended treatment. The death rate was found to be as high as 40% and 69% in children with severe sepsis and septic shock respectively with co-morbidities such as severe malnutrition.
2. Knowledge gap: The conventional management of SAM children with features of severe sepsis recommended by WHO include administration of boluses of isotonic saline followed by blood transfusion in unresponsive cases with septic shock. However, a recent African study reported significantly higher mortality among children with features of severe sepsis when they were treated with boluses. To date, no study has evaluated systematically the effects of inotrope or vasopressor or blood transfusion in children with dehydrating diarrhea (for example, in cholera) and SAM having shock and unresponsive to WHO standard fluid therapy.
3. Relevance: If this randomized trial signifies survival benefit from a blood transfusion, inotrope or vasopressor in the management of fluid refractory shock in children with severe acute malnutrition and cholera or other dehydrating diarrheas, then this approach would be a good candidate for implementation in the management of such children especially in developing countries

Hypothesis: We hypothesize that the death rates will be significantly lower in children with SAM or severe underweight, dehydrating diarrhea and fluid refractory shock who will be treated with blood transfusion and adrenaline compared to blood transfusion and dopamine, after treatment failure with WHO standard bolus intravenous fluid therapy.

Objectives: To reduce mortality of the SAM or severely underweight children presenting with diarrhea and fluid refractory shock who will receive WHO standard fluid therapy followed by blood transfusion with either dopamine or adrenaline.

Methods: This will be a randomized, two-arm, controlled, non-masked clinical trial in children 1- 59 months old with SAM or severely underweight and fluid refractory shock. It will compare the efficacy of WHO-recommended fluid resuscitation followed by blood transfusion and dopamine versus blood transfusion and adrenaline. Children in both groups will also receive inj hydrocortisone. After parental written informed consent, children, in addition to usual supportive care, will be allocated to the study interventions following randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Children of either sex with acute malnutrition and diarrhea
2. Age: 1-59 months
3. Children with cerebral palsy (CP) and/or developmental delay, Down Syndrome with or without heart diseases
4. Fluid refractory shock
5. Consent from the caregivers/parents

Exclusion Criteria:

1. Having a rare blood group (Rh negative blood groups provided that donor is not available)
2. A child requiring cardio-pulmonary resuscitation during screening or having gasping respiration

Ages: 1 Month to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Case fatality rate | 28 days (± 3 days)
  Number of mortalities among acutely malnourished children presenting with diarrhea and fluid refractory shock who would receive WHO standard fluid therapy followed by blood transfusion with either dopamine or adrenaline.

SECONDARY OUTCOMES:
Treatment failure rates | Through study completion, an average of 7 days
  Number of children where we failed to achieve the goal of resuscitation after starting any one of the interventions
Need for mechanical ventilation | Through study completion, an average of 7 days
  Number of children who would require mechanical ventilation
Heart failure | Through study completion, an average of 7 days
  Number of children who developed heart failure. Heart failure will be assessed on the basis of - age-specific tachypnea, tachycardia, enlarged tender liver, pedal edema, basal crackles and/or gallop and response to furosemide (combination of findings).
Length of ICU stay | Through study completion, an average of 7 days
  Time a child stays in ICU
Time-to-achieve recovery | 3-4 hours
  Required times (minutes) for resuscitation of a child after randomization to a specific arms
Left ventricular function of the study participants | Through study completion, an average of 7 days
  Evaluation of left ventricular function (hyperdynamic or normal) by cardiac USG at enrollment, at time of heart failure (if any)
Right ventricular function of the study participants | Through study completion, an average of 7 days
  Evaluation of right ventricular function (hyperdynamic or normal) by cardiac ultrasound at enrollment, at time of heart failure (if any)
Inferior vena cava collapsibility of the study participants | Through study completion, an average of 7 days
  Evaluation of Inferior vena cava collapsibility by cardiac ultrasound at enrollment, at time of heart failure (if any)
Length of hospital stay | variable (days to months)
  Time a child stays in the hospital
Mean arterial pressure (MAP) stabilization at 48 hours | 48 hours from the point of inclusion in the study
  Number of children whose MAP was stabilized at 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tahmeed Ahmed, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chisti MJ, Pietroni MA, Smith JH, Bardhan PK, Salam MA. Predictors of death in under-five children with diarrhoea admitted to a critical care ward in an urban hospital in Bangladesh. Acta Paediatr. 2011 Dec;100(12):e275-9. doi: 10.1111/j.1651-2227.2011.02368.x. Epub 2011 Jun 21. PMID 21627690
- [Background] Sarmin M, Ahmed T, Bardhan PK, Chisti MJ. Specialist hospital study shows that septic shock and drowsiness predict mortality in children under five with diarrhoea. Acta Paediatr. 2014 Jul;103(7):e306-11. doi: 10.1111/apa.12640. Epub 2014 Apr 11. PMID 24661049
- [Background] Ahmed T, Ali M, Ullah MM, Choudhury IA, Haque ME, Salam MA, Rabbani GH, Suskind RM, Fuchs GJ. Mortality in severely malnourished children with diarrhoea and use of a standardised management protocol. Lancet. 1999 Jun 5;353(9168):1919-22. doi: 10.1016/S0140-6736(98)07499-6. PMID 10371570
- [Background] Chisti MJ, Salam MA, Bardhan PK, Faruque AS, Shahid AS, Shahunja KM, Das SK, Hossain MI, Ahmed T. Severe Sepsis in Severely Malnourished Young Bangladeshi Children with Pneumonia: A Retrospective Case Control Study. PLoS One. 2015 Oct 6;10(10):e0139966. doi: 10.1371/journal.pone.0139966. eCollection 2015. PMID 26440279
- [Background] Sarker AR, Sultana M, Mahumud RA, Ali N, Huda TM, Salim Uzzaman M, Haider S, Rahman H, Islam Z, Khan JAM, Van Der Meer R, Morton A. Economic costs of hospitalized diarrheal disease in Bangladesh: a societal perspective. Glob Health Res Policy. 2018 Jan 5;3:1. doi: 10.1186/s41256-017-0056-5. eCollection 2018. PMID 29318195
- [Background] Guerrant RL, Schorling JB, McAuliffe JF, de Souza MA. Diarrhea as a cause and an effect of malnutrition: diarrhea prevents catch-up growth and malnutrition increases diarrhea frequency and duration. Am J Trop Med Hyg. 1992 Jul;47(1 Pt 2):28-35. doi: 10.4269/ajtmh.1992.47.28. PMID 1632474
- [Background] Pocket Book of Hospital Care for Children: Guidelines for the Management of Common Childhood Illnesses. 2nd edition. Geneva: World Health Organization; 2013. Available from http://www.ncbi.nlm.nih.gov/books/NBK154447/ PMID 24006557
- [Background] Chisti MJ, Saha S, Roy CN, Salam MA. Predictors of bacteremia in infants with diarrhea and systemic inflammatory response syndrome attending an urban diarrheal treatment center in a developing country. Pediatr Crit Care Med. 2010 Jan;11(1):92-7. doi: 10.1097/PCC.0b013e3181b063e1. PMID 19593244
- [Background] Ranjit S, Aram G, Kissoon N, Ali MK, Natraj R, Shresti S, Jayakumar I, Gandhi D. Multimodal monitoring for hemodynamic categorization and management of pediatric septic shock: a pilot observational study*. Pediatr Crit Care Med. 2014 Jan;15(1):e17-26. doi: 10.1097/PCC.0b013e3182a5589c. PMID 24196006
- [Background] Davis AL, Carcillo JA, Aneja RK, Deymann AJ, Lin JC, Nguyen TC, Okhuysen-Cawley RS, Relvas MS, Rozenfeld RA, Skippen PW, Stojadinovic BJ, Williams EA, Yeh TS, Balamuth F, Brierley J, de Caen AR, Cheifetz IM, Choong K, Conway E Jr, Cornell T, Doctor A, Dugas MA, Feldman JD, Fitzgerald JC, Flori HR, Fortenberry JD, Graciano AL, Greenwald BM, Hall MW, Han YY, Hernan LJ, Irazuzta JE, Iselin E, van der Jagt EW, Jeffries HE, Kache S, Katyal C, Kissoon N, Kon AA, Kutko MC, MacLaren G, Maul T, Mehta R, Odetola F, Parbuoni K, Paul R, Peters MJ, Ranjit S, Reuter-Rice KE, Schnitzler EJ, Scott HF, Torres A Jr, Weingarten-Arams J, Weiss SL, Zimmerman JJ, Zuckerberg AL. American College of Critical Care Medicine Clinical Practice Parameters for Hemodynamic Support of Pediatric and Neonatal Septic Shock. Crit Care Med. 2017 Jun;45(6):1061-1093. doi: 10.1097/CCM.0000000000002425. PMID 28509730
- [Background] Maitland K, Kiguli S, Opoka RO, Engoru C, Olupot-Olupot P, Akech SO, Nyeko R, Mtove G, Reyburn H, Lang T, Brent B, Evans JA, Tibenderana JK, Crawley J, Russell EC, Levin M, Babiker AG, Gibb DM; FEAST Trial Group. Mortality after fluid bolus in African children with severe infection. N Engl J Med. 2011 Jun 30;364(26):2483-95. doi: 10.1056/NEJMoa1101549. Epub 2011 May 26. PMID 21615299
- [Background] Seri I, Abbasi S, Wood DC, Gerdes JS. Regional hemodynamic effects of dopamine in the sick preterm neonate. J Pediatr. 1998 Dec;133(6):728-34. doi: 10.1016/s0022-3476(98)70141-6. PMID 9842034
- [Background] Maitland K, George EC, Evans JA, Kiguli S, Olupot-Olupot P, Akech SO, Opoka RO, Engoru C, Nyeko R, Mtove G, Reyburn H, Brent B, Nteziyaremye J, Mpoya A, Prevatt N, Dambisya CM, Semakula D, Ddungu A, Okuuny V, Wokulira R, Timbwa M, Otii B, Levin M, Crawley J, Babiker AG, Gibb DM; FEAST trial group. Exploring mechanisms of excess mortality with early fluid resuscitation: insights from the FEAST trial. BMC Med. 2013 Mar 14;11:68. doi: 10.1186/1741-7015-11-68. PMID 23496872
- [Background] Phornphatkul C, Pongprot Y, Suskind R, George V, Fuchs G. Cardiac function in malnourished children. Clin Pediatr (Phila). 1994 Mar;33(3):147-54. doi: 10.1177/000992289403300304. PMID 8194289
- [Background] Ventura AM, Shieh HH, Bousso A, Goes PF, de Cassia F O Fernandes I, de Souza DC, Paulo RL, Chagas F, Gilio AE. Double-Blind Prospective Randomized Controlled Trial of Dopamine Versus Epinephrine as First-Line Vasoactive Drugs in Pediatric Septic Shock. Crit Care Med. 2015 Nov;43(11):2292-302. doi: 10.1097/CCM.0000000000001260. PMID 26323041
- [Background] Ramaswamy KN, Singhi S, Jayashree M, Bansal A, Nallasamy K. Double-Blind Randomized Clinical Trial Comparing Dopamine and Epinephrine in Pediatric Fluid-Refractory Hypotensive Septic Shock. Pediatr Crit Care Med. 2016 Nov;17(11):e502-e512. doi: 10.1097/PCC.0000000000000954. PMID 27673385
- [Background] Weiss SL, Peters MJ, Alhazzani W, Agus MSD, Flori HR, Inwald DP, Nadel S, Schlapbach LJ, Tasker RC, Argent AC, Brierley J, Carcillo J, Carrol ED, Carroll CL, Cheifetz IM, Choong K, Cies JJ, Cruz AT, De Luca D, Deep A, Faust SN, De Oliveira CF, Hall MW, Ishimine P, Javouhey E, Joosten KFM, Joshi P, Karam O, Kneyber MCJ, Lemson J, MacLaren G, Mehta NM, Moller MH, Newth CJL, Nguyen TC, Nishisaki A, Nunnally ME, Parker MM, Paul RM, Randolph AG, Ranjit S, Romer LH, Scott HF, Tume LN, Verger JT, Williams EA, Wolf J, Wong HR, Zimmerman JJ, Kissoon N, Tissieres P. Surviving Sepsis Campaign International Guidelines for the Management of Septic Shock and Sepsis-Associated Organ Dysfunction in Children. Pediatr Crit Care Med. 2020 Feb;21(2):e52-e106. doi: 10.1097/PCC.0000000000002198. PMID 32032273
- [Background] Sun JT. New Advances in Emergency Ultrasound Protocols for Shock. J Med Ultrasound. 2017 Oct-Dec;25(4):191-194. doi: 10.1016/j.jmu.2017.09.005. Epub 2017 Dec 6. No abstract available. PMID 30065491
- [Background] Sekiguchi H, Harada Y, Villarraga HR, Mankad SV, Gajic O. Focused cardiac ultrasound in the early resuscitation of severe sepsis and septic shock: a prospective pilot study. J Anesth. 2017 Aug;31(4):487-493. doi: 10.1007/s00540-017-2312-8. Epub 2017 Jan 31. PMID 28144779
- [Background] McQuilten ZK, Cooper DJ. Age of Red Blood Cells for Transfusion in Critically Ill Pediatric Patients. JAMA. 2019 Dec 10;322(22):2175-2176. doi: 10.1001/jama.2019.17476. No abstract available. PMID 31821418
- [Background] Tiwari AK, Aggarwal G, Dara RC, Arora D, Gupta GK, Raina V. First Indian study to establish safety of immediate-spin crossmatch for red blood cell transfusion in antibody screen-negative recipients. Asian J Transfus Sci. 2017 Jan-Jun;11(1):40-44. doi: 10.4103/0973-6247.200774. PMID 28316439
- [Background] AABB. Technical Manual. 19th ed. Fung MK, Eder AF, Spitalnik SL, Westhoff CM, editors. United States.
- [Background] Green REB, Klostermann DA. The Antiglobulin Test. In: Harmening D, editor. Modern Blood Banking & Transfusion Practices. 6th ed. Philadelphia: F.A. Davis. p. 107-10.
- [Derived] Sarmin M, Shaly NJ, Sultana T, Tariqujjaman M, Shikha SS, Mariam N, Jeorge DH, Tabassum M, Nahar B, Afroze F, Shahrin L, Hossain MI, Alam B, Faruque ASG, Islam MM, Osmany DMF, Ahmed CM, Manji K, Kissoon N, Chisti MJ, Ahmed T. Efficacy of dopamine, epinephrine and blood transfusion for treatment of fluid refractory shock in children with severe acute malnutrition or severe underweight and cholera or other dehydrating diarrhoeas: protocol for a randomised controlled clinical trial. BMJ Open. 2023 Apr 12;13(4):e068660. doi: 10.1136/bmjopen-2022-068660. PMID 37045565